CLINICAL TRIAL: NCT04275856
Title: Etiology, Incidence and Survival of Pediatric Out-of-hospital Cardiac Arrests: a Four-year Danish Analysis
Acronym: Child-OHCA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: Odense University Hospital (Other); Aalborg University Hospital (Other); TrygFonden, Denmark (Industry)
Responsible Party: Sponsor
Other Study IDs: Child-OHCA
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Pediatric Disorder; Cardiopulmonary Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: OHCA is a rare condition for children and young adults. Overall incidence rates are reported as 3.3-5.97 per 100.000 inhabitants. Previous studies from different data sources have identified a diverse and slightly incompatible etiologies. The purpose of this investigation was to analyze presumed etiologies of pediatric OHCA and report incident and survival rates. Further the investigators wish to present central characteristics of pediatric OHCA in Denmark.

Methods: Data will be collected from the verified 2016-2019 Danish OHCA register. Inclusion criteria were age ≤ 16 years at the time of the event. All included EMS reports will read by two authors [MGH and TWJ] and the presumed reversible cause assigned to each case. Incidence rates per 100.000 citizens, survival rates to hospital, initial rhythm, use of AED by laypersons, EMS treatment and presumed etiology are reported.

To test feasibility a study was conducted in 2018, on the 56 verified cases of children with OHCA was reported in the capital region of Denmark in 2016-2018 (among 1.8 million inhabitants). Incident rates were 0.83-1.34 per 100.000 inhabitants per year. Preliminary data show survival to hospital was 46% which was markedly higher than the adult population (28%, p = 0.002).

The most common cause of OHCA was hypoxia (50%) followed by trauma/hypovolemia (14%) and others (7%). Approximately 23% did not present with an apparent etiology. Hereditary disorders as the primary cause was noted in 7% of the cases.

The conclusion from the feasibility study is that the study is possible and that a reasonable proportion of pediatric OHCA can be analyzed from EMS medical reports.

Expected outcome:

Variables included in the study: age, gender, initial rhythm, etiology of cardiac arrest, event location, observation of occurrence, cardio-pulmonary-resuscitation (CPR), defibrillation and use automatic external defibrillators (AEDs), EMS-response time, hospitalization, return-of-spontaneous-circulation (ROSC), state at hospital admission, 30-day survival, airway management and use of epinephrine. See the dedicated study protocol for an extended description of the variables and associated analyses.

DETAILED DESCRIPTION:
Background In 2016 the Danish Emergency Medical Services (EMS) introduced a nationwide electronic medical reporting system. This provided new possibilities for exploring many of the aspects surrounding the daily practice the EMS, including information on selective subgroups of cardiac arrest patients. The Danish out-of-hospital cardiac arrests (OHCA) registry is based on electronic EMS reports together with a strenuous manual validation process. The product is a solid base for identification and verification of OHCA. Whenever a cardiac arrest is identified, EMS medical reports can be accessed supplying information on the background, observations and treatments that can be extracted systematically. The gain of insight from this process, provide us with the possibility to explore several novel aspects of pediatric OHCA.

OHCA is a rare event in pediatric populations with varying reports of incidence rates, ranging from 3.3 to 19.7 per 100.000 person years. Most studies, however, are centered around an incidence rate of about 8-9/100.000 person years. Generally, increased incidence rates are reported for infants compared to older children, and discrepancies in the overall incidence rates could partly be explained by different age-caps when defining the pediatric population. These inconsistencies unfortunately underline a general trend in pediatric OHCA studies, with different term definitions and data validation obscuring the overall overview and complicating more in-depth aggregate analyses. This calls for more high-quality data sources, including data validation, and a more strict adherence to standardized reporting templates such as the Utstein style for pediatric advanced life support (PALS).

Unquestionably, pediatric settings of cardiac arrest embarks an inherent urge to perform beyond ones supreme, but though discrepancies exist, overall survival is reported to be less than 11%, with 30-day survival ranging from 8.1% to 11%, and survival until hospital discharge ranging from 2% to 10.9%. This leads to a potential for improvement, which requires first and foremost clarification of the most obvious causes.

The etiology of OHCA is often categorized by cardiac or non-cardiac etiology as an object of prevention and post-mortem determination. However, OHCA in children are less likely to be a primary cardiac event. When the focus is solely on increasing survival, reversible causes is more often the focus and is labelled a key component of adult advanced resuscitation algorithms. The most commonly used denomination for reversible causes to consider during advanced life support is "H's" (Hypoxia, Hypovolemia, Hydrogen ion (acidosis), Hypo-/hyperkalemia and Hypothermia) and "T's"(Toxins, Tamponade cardiac, Tension pneumothorax, Thrombosis, pulmonary and Thrombosis coronary). Likewise, PALS operate in "H's" and "T's", and more often than not, prescribe a primary focus on hypoxia as the most prominent reversible cause.

The investigators speculate that the EMS medical reports provide new and central information about etiology and, perhaps more central to survival, reversible causes of pediatric OHCA.

Aim The purpose of this analysis is to describe the incidence, presumed etiology and survival-rates for pediatric OHCA within a four-year period in a Danish setting.

Methods The study is a registry-based follow-up, including prehospital medical record registrations of pediatric EMS patients in Denmark in 2016, 2017, 2018 and 2019 with cardiac arrest.

Data source:

This analysis will be based on data from the national verified Danish OHCA registry. In, Denmark all cases of OHCA with resuscitative attempts are immediately followed up with recording of specific data, including EMS reports, aimed at the registry. In 2016 the registry became electronic, as one central database enabling an easier approach to research on OHCA. The registry contains approximately 5.400 registrations of OHCA annually. These composed of active entries, as well as advanced text searches of prehospital patient charts maximizing the likelihood of identifying and collecting all possible cardiac arrests. In a large validation process, all identified cases are read through manually by an external verification team, ensuring a high standard of data quality. During this process, several additional data sources is coupled with each registered OHCA, notably survival, initiation of bystander CPR and actions from EMS personnel.

Identification of pediatric cardiac arrests:

The external verification team indirectly mark cases as pediatric, whenever a subject is less than 16 years of age at the time of the event. This together with age derived from individual personal identification numbers is used to identify all pediatric cases. All Danish citizens is provided with a unique personal identification number at birth, containing the individuals date-of-birth. Subjects reported as unquestionably deceased (late signs of death) at EMS arrival will be excluded.

Identification of presumed causes:

Three individual raters [MGH, TWJ and NB] will independently review all cases for an assessment of the suspected cause of arrest and assign a presumed reversible cause based on "H's" and "T's" alongside a free-text description for justification. Disagreement will be resolved by third party members [HCC, SM or FL]. If a case does not present with any obvious information indicating a reversible cause or with several competing reversible causations, the cases will be denoted as "NA" and "Inconclusive" respectively. If a case is obviously a result of a chronic disease and no reversible causality was possible the case will be noted "non-reversible".

Variables included:

* Age: Age will be defined as the subject age at the time of the event. Subjects will be stratified into four age-groups, including; infants (<1 years of age), pre-school children (1-5 years of age), school children (6-12 years of age) and teenagers (>12 years of age).
* Gender: Gender will be defined as either male, female or undetermined, and derived from personal identification numbers. In the expected minority of cases without a number, gender will, as far as possible, be defined based on EMS-charts.
* Initial rhythm: The initial rhythm will be defined as the first rhythm observed by EMS personnel, and categorized as either shockable, non-shockable (asystole), non-shockable (other) and undetermined.
* Etiology of cardiac arrest: Presumed etiology will be categorized as either reversible (including a subcategorization into the 4H's and 4T's) and non-reversible. Further, the investigators aim to categorize the preceding event, stratifying this into either; a medical cause, trauma, drug overdose, drowning, asphyxia, sports-related or suicide.
* Event location: This will be classified as either; private home, public space, outdoor nature or other.
* Observation of occurrence: Arrests will be classified as either unwitnessed, bystander witnessed or EMS-witnessed.
* Cardio-pulmonary-resuscitation (CPR): CPR will include bystander initiated and EMS treatment with CPR.
* Defibrillation and use automatic external defibrillators (AEDs): Defibrillation will include defibrillation by bystanders and/or EMS personnel, including the use of publicly available AEDs that have analyzed the rhythm without delivering shocks.
* EMS-response time: This will include the time between a dispatcher receiving the emergency call and the arrival of the first EMS-personnel.
* Hospitalization: This will be categorized as either; transported to hospital or declared dead by EMS-personnel.
* Return-of-spontaneous-circulation (ROSC): ROSC will be defined as cases achieving ROSC anytime between recognition of the event and termination (defined as either hospital admission og declaration of death by EMS-personnel).
* State at hospital admission: The investigators will define the case state on arrival at the hospital as either; ROSC or ongoing CPR.
* Survival: Survival will be defined as ROSC at the time of hospital admission, further the investigators will include rates for 30-day survival derived with data from the National Patient Registry.
* Airway management: The investigators aim to describe the airway maneuvers performed on each case by listing the use of nasopharyngeal airways, oropharyngeal airways, endo-tracheal intubation, supraglottic airways and isolated bag-valve-mask ventilation.
* Use of epinephrine: This will include a binary (yes/no) variable based upon the potential administration of epinephrine for each case.

Analysis and presentation of data:

The primary aim of this study is to provide a descriptive analysis of the reversible causes (H's and T's) in a Danish nationwide setting of pediatric OHCA. The secondary goal is to provide updated annual incidence- and survival rates. Descriptive statistics will include the variables listed above with a denotation of the absolute numbers with percentages and stratified in the specified age-groups. Comparative analyses, addressing between age-group differences, will be performed using non-parametric statistics. The data will be pseudo-anonymized all analyses will be performed on an aggregated nationwide level. The primary outcome is ROSC at hospital admission, in relation to reversible causes and age-groups. The secondary outcome is 30-day survival in relation to reversible causes. Final outcomes will be compared to a control-group of adult OHCA with an aim to quantify differences in survival including influencing variables.

Pilot study:

Prior to this study, the investigators initiated a pilot project based on available data (from 2016-2019) from the capital region of Denmark within the verified Danish OHCA registry. The aim was to investigate the feasibility of the proposed methods. The investigators identified 56 cases and were able to deduct a presumed cause in 73% of cases. Reasonably amounts of information was attainable from exploration of the prehospital EMS-charts. The other Danish regions will provide data with a similar setup, and hence the investigators expect the presumed methods to be feasible at a nationwide level.

Perspective The descriptive part of this study will provide updated realistic numbers on pediatric OHCA from a thoroughly reviewed, high-quality database. In addition, a review for reversible causes will contribute to an understanding of the extent of cardiac arrests where focus should be extended to involve more than hypoxia, including associated survival rates.

List of abbreviations EMS: Emergency Medical Service OHCA: Out-of-hospital cardiac arrest PALS: Pediatric Advanced Life Support CPR: Cardio-pulmonary resuscitation AED: Automated External Defibrillation ROSC: Return of spontaneous circulation GDRP: General Data Protection Regulation

ELIGIBILITY:
Inclusion Criteria:

* All out-of-hospital cardiac arrests victim from 0-16 year of age.
* The external verification team indirectly mark cases as pediatric, whenever a subject is less than 16 years of age at the time of the event. This together with age derived from individual personal identification numbers is used to identify all pediatric cases. All Danish citizens is provided with a unique personal identification number at birth, containing the individuals date-of-birth.

Exclusion Criteria:

* Subjects reported as unquestionably deceased (late signs of death) at EMS arrival will be excluded.

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The external verification team indirectly mark cases as pediatric, whenever a subject is less than 16 years of age at the time of the event. This together with age derived from individual personal identification numbers is used to identify all pediatric cases. All Danish citizens is provided with a unique personal identification number at birth, containing the individuals date-of-birth.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Return-of-spontaneous-circulation (ROSC) | Through study completion, an average of 1 year
  ROSC will be defined as cases achieving ROSC anytime between recognition of the event and termination (defined as either hospital admission og declaration of death by EMS-personnel).
State at hospital admission | Through study completion, an average of 1 year
  The investigators will define the case state on arrival at the hospital as either; ROSC or ongoing CPR.
30-day Survival | Through study completion, an average of 1 year
  Survival will be defined as ROSC at the time of hospital admission. Further the investigators will include rates for 30-day survival derived with data from the National Patient Registry.
Etiology of cardiac arrest | Through study completion, an average of 1 year
  Presumed etiology will be categorized as either reversible (including a subcategorization into the 4H's and 4T's) and non-reversible. Further, the investigators aim to categorise the preceding event, stratifying this into either; a medical cause, trauma, drug overdose, drowning, asphyxia, sports-related or suicide.
Incidence rate | Through study completion, an average of 1 year
  Incidence rate of paediatric out-of-hospital cardiac arrest per 100.000 citizens and equivalent measures for age specific subgroups

OTHER OUTCOMES:
Airway management | Through study completion, an average of 1 year
  The investigators aim to describe the airway maneuvers performed on each case by listing the use of nasopharyngeal airways, oropharyngeal airways, endo-tracheal intubation, supraglottic airways and isolated bag-valve-mask ventilation.
Use of epinephrine | Through study completion, an average of 1 year
  This will include a binary (yes/no) variable based upon the potential administration of epinephrine for each case.
Defibrillation and use automatic external defibrillators (AEDs) | Through study completion, an average of 1 year
  Defibrillation will include defibrillation by bystanders and/or EMS personnel, including the use of publicly available AEDs that have analyzed the rhythm without delivering shocks.
Initial rhythm | Through study completion, an average of 1 year
  The initial rhythm will be defined as the first rhythm observed by EMS personnel, and categorized as either shockable, non-shockable (asystole), non-shockable (other) and undetermined.

CONTACTS AND LOCATIONS:
Overall Officials: Freddy K Lippert, MD, Ass. Professor, Study Chair — Copenhagen Emergency Medical Services
Locations (1):
- Copenhagen Emergency Medical Services, Copenhagen, Denmark

REFERENCES:
- [Background] Lindskou TA, Mikkelsen S, Christensen EF, Hansen PA, Jorgensen G, Hendriksen OM, Kirkegaard H, Berlac PA, Sovso MB. The Danish prehospital emergency healthcare system and research possibilities. Scand J Trauma Resusc Emerg Med. 2019 Nov 4;27(1):100. doi: 10.1186/s13049-019-0676-5. PMID 31684982
- [Background] Rajan S, Wissenberg M, Folke F, Hansen CM, Lippert FK, Weeke P, Karlsson L, Sondergaard KB, Kragholm K, Christensen EF, Nielsen SL, Kober L, Gislason GH, Torp-Pedersen C. Out-of-hospital cardiac arrests in children and adolescents: incidences, outcomes, and household socioeconomic status. Resuscitation. 2015 Mar;88:12-9. doi: 10.1016/j.resuscitation.2014.11.025. Epub 2014 Dec 10. PMID 25500748
- [Background] Ong ME, Stiell I, Osmond MH, Nesbitt L, Gerein R, Campbell S, McLellan B; OPALS Study Group. Etiology of pediatric out-of-hospital cardiac arrest by coroner's diagnosis. Resuscitation. 2006 Mar;68(3):335-42. doi: 10.1016/j.resuscitation.2005.05.026. Epub 2006 Feb 7. PMID 16455177
- [Background] Sirbaugh PE, Pepe PE, Shook JE, Kimball KT, Goldman MJ, Ward MA, Mann DM. A prospective, population-based study of the demographics, epidemiology, management, and outcome of out-of-hospital pediatric cardiopulmonary arrest. Ann Emerg Med. 1999 Feb;33(2):174-84. doi: 10.1016/s0196-0644(99)70391-4. PMID 9922413
- [Background] Kuisma M, Suominen P, Korpela R. Paediatric out-of-hospital cardiac arrests--epidemiology and outcome. Resuscitation. 1995 Oct;30(2):141-50. doi: 10.1016/0300-9572(95)00888-z. PMID 8560103
- [Background] Gerein RB, Osmond MH, Stiell IG, Nesbitt LP, Burns S; OPALS Study Group. What are the etiology and epidemiology of out-of-hospital pediatric cardiopulmonary arrest in Ontario, Canada? Acad Emerg Med. 2006 Jun;13(6):653-8. doi: 10.1197/j.aem.2005.12.025. Epub 2006 May 2. PMID 16670256
- [Background] Atkins DL, Everson-Stewart S, Sears GK, Daya M, Osmond MH, Warden CR, Berg RA; Resuscitation Outcomes Consortium Investigators. Epidemiology and outcomes from out-of-hospital cardiac arrest in children: the Resuscitation Outcomes Consortium Epistry-Cardiac Arrest. Circulation. 2009 Mar 24;119(11):1484-91. doi: 10.1161/CIRCULATIONAHA.108.802678. Epub 2009 Mar 9. PMID 19273724
- [Background] Bardai A, Berdowski J, van der Werf C, Blom MT, Ceelen M, van Langen IM, Tijssen JG, Wilde AA, Koster RW, Tan HL. Incidence, causes, and outcomes of out-of-hospital cardiac arrest in children. A comprehensive, prospective, population-based study in the Netherlands. J Am Coll Cardiol. 2011 May 3;57(18):1822-8. doi: 10.1016/j.jacc.2010.11.054. PMID 21527156
- [Background] Zaritsky A, Nadkarni V, Hazinski MF, Foltin G, Quan L, Wright J, Fiser D, Zideman D, O'Malley P, Chameides L. Recommended guidelines for uniform reporting of pediatric advanced life support: the pediatric Utstein Style. A statement for healthcare professionals from a task force of the American Academy of Pediatrics, the American Heart Association, and the European Resuscitation Council. Writing Group. Circulation. 1995 Oct 1;92(7):2006-20. doi: 10.1161/01.cir.92.7.2006. PMID 7671387
- [Background] Akahane M, Tanabe S, Ogawa T, Koike S, Horiguchi H, Yasunaga H, Imamura T. Characteristics and outcomes of pediatric out-of-hospital cardiac arrest by scholastic age category. Pediatr Crit Care Med. 2013 Feb;14(2):130-6. doi: 10.1097/PCC.0b013e31827129b3. PMID 23314182
- [Background] Fukuda T, Kondo Y, Hayashida K, Sekiguchi H, Kukita I. Time to epinephrine and survival after paediatric out-of-hospital cardiac arrest. Eur Heart J Cardiovasc Pharmacother. 2018 Jul 1;4(3):144-151. doi: 10.1093/ehjcvp/pvx023. PMID 29036580
- [Background] Hansen ML, Lin A, Eriksson C, Daya M, McNally B, Fu R, Yanez D, Zive D, Newgard C; CARES surveillance group. A comparison of pediatric airway management techniques during out-of-hospital cardiac arrest using the CARES database. Resuscitation. 2017 Nov;120:51-56. doi: 10.1016/j.resuscitation.2017.08.015. Epub 2017 Aug 22. PMID 28838781
- [Background] Jayaram N, McNally B, Tang F, Chan PS. Survival After Out-of-Hospital Cardiac Arrest in Children. J Am Heart Assoc. 2015 Oct 8;4(10):e002122. doi: 10.1161/JAHA.115.002122. PMID 26450118
- [Background] Deasy C, Bernard SA, Cameron P, Jaison A, Smith K, Harriss L, Walker T, Masci K, Tibballs J. Epidemiology of paediatric out-of-hospital cardiac arrest in Melbourne, Australia. Resuscitation. 2010 Sep;81(9):1095-100. doi: 10.1016/j.resuscitation.2010.04.029. Epub 2010 Jun 2. PMID 20627518
- [Background] Tirkkonen J, Hellevuo H, Olkkola KT, Hoppu S. Aetiology of in-hospital cardiac arrest on general wards. Resuscitation. 2016 Oct;107:19-24. doi: 10.1016/j.resuscitation.2016.07.007. Epub 2016 Aug 1. PMID 27492850
- [Background] Vega RM EP. Cardiopulmonary Arrest - PubMed - NCBI [Internet]. [cited 2020 Feb 7]. Available from: https://www.ncbi.nlm.nih.gov/pubmed/?term=Cardiopulmonary+Arrest+Vega+RM
- [Background] Andersen LW, Holmberg MJ, Berg KM, Donnino MW, Granfeldt A. In-Hospital Cardiac Arrest: A Review. JAMA. 2019 Mar 26;321(12):1200-1210. doi: 10.1001/jama.2019.1696. PMID 30912843
- [Background] Soar J, Nolan JP, Bottiger BW, Perkins GD, Lott C, Carli P, Pellis T, Sandroni C, Skrifvars MB, Smith GB, Sunde K, Deakin CD; Adult advanced life support section Collaborators. European Resuscitation Council Guidelines for Resuscitation 2015: Section 3. Adult advanced life support. Resuscitation. 2015 Oct;95:100-47. doi: 10.1016/j.resuscitation.2015.07.016. No abstract available. PMID 26477701
- [Background] Durila M. Reversible causes of cardiac arrest 4 "Ts" and 4 "Hs" can be easily diagnosed and remembered following general ABC rule, Motol University Hospital approach. Resuscitation. 2018 May;126:e7. doi: 10.1016/j.resuscitation.2018.03.013. Epub 2018 Mar 12. No abstract available. PMID 29545140
- [Background] Field RA. From changing four tyres to recalling the four H's and T's - Can the pit crew model work for in-hospital cardiac arrest? Resuscitation. 2019 Oct;143:212-213. doi: 10.1016/j.resuscitation.2019.08.002. Epub 2019 Aug 29. No abstract available. PMID 31473263
- [Background] Neumar RW, Otto CW, Link MS, Kronick SL, Shuster M, Callaway CW, Kudenchuk PJ, Ornato JP, McNally B, Silvers SM, Passman RS, White RD, Hess EP, Tang W, Davis D, Sinz E, Morrison LJ. Part 8: adult advanced cardiovascular life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S729-67. doi: 10.1161/CIRCULATIONAHA.110.970988. PMID 20956224
- [Background] Duff JP, Topjian A, Berg MD, Chan M, Haskell SE, Joyner BL Jr, Lasa JJ, Ley SJ, Raymond TT, Sutton RM, Hazinski MF, Atkins DL. 2018 American Heart Association Focused Update on Pediatric Advanced Life Support: An Update to the American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2018 Dec 4;138(23):e731-e739. doi: 10.1161/CIR.0000000000000612. PMID 30571264
- [Background] Hunt EA, Duval-Arnould JM, Bembea MM, Raymond T, Calhoun A, Atkins DL, Berg RA, Nadkarni VM, Donnino M, Andersen LW; American Heart Association's Get With The Guidelines-Resuscitation Investigators. Association Between Time to Defibrillation and Survival in Pediatric In-Hospital Cardiac Arrest With a First Documented Shockable Rhythm. JAMA Netw Open. 2018 Sep 7;1(5):e182643. doi: 10.1001/jamanetworkopen.2018.2643. PMID 30646171